CLINICAL TRIAL: NCT05477602
Title: The Automated Calculation of AF Cycle Length and Complexity Using a Novel EP Recording System (The CathVision ECGenius System)
Brief Title: The Automated Calculation of AF Cycle Length and Complexity Using a Novel EP Recording System
Status: Completed | Type: Observational
Sponsor: CathVision ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: CVAR-00002-A
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: electrophysiology; cardiac ablation; persistent atrial fibrillation; cycle length
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac Ablation for the treatment of persistent Atrial Fibrillation — Patients undergoing cardiac ablation for the treatment of persistent atrial fibrillation
  Other Names: Persistent AF Ablation

SUMMARY:
Collect electrophysiological data during atrial fibrillation (AF) ablation procedures to assess the performance of a Signal Complexity Visualization algorithm designed to be integrated into the CathVision ECGenius® System.

DETAILED DESCRIPTION:
A prospective, single-center, feasibility study using the CathVision ECGenius® system and a Signal Complexity Visualization Algorithm during radiofrequency (RF) ablation procedures to treat persistent AF.

Subjects with persistent AF who are indicated to undergo a routine-practice RF ablation may be enrolled in the Study. Intracardiac signals will be passively recorded using the investigational CathVision ECGenius® System in parallel with a commercial (CE Approved) EP recording system. The investigational device will not be used for direct clinical care decisions or therapy.

The validation of the Signal Complexity Visualization Algorithm will be performed offline and retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing RF ablation indicated by the investigator for the treatment of persistent atrial fibrillation.
* Male or non-pregnant female aged ≥ 21 years.
* Able and willing to provide written informed consent prior to any clinical investigation related procedure.

Exclusion Criteria:

* Current participation in another investigational drug or device study that interferes with this study.
* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
* Life expectancy less than 12 month, in the opinion of the Investigator.
* Subjects who, in the opinion of the investigator, are not candidates for this study.
* Subjects who, in the opinion of the investigator, are considered part of any vulnerable population.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for a cardiac ablation for the treatment of persistent atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- OLV Aalst, Aalst, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Full Cohort: All patients recruited
Period: Overall Study
Arm/Group | Full Cohort
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1 patient did not meet the eligibility criteria after screening
Groups:
- Full Cohort: All 21 patients in the PPT group
Arm/Group | Full Cohort
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.29 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kg] | 81.57 (17.71)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 138.48 (21.18)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 86.33 (12.59)
Heart Rate [Mean (Standard Deviation); unit: BPM] | 78.9 (19.54)
Respiratory Rate [Mean (Standard Deviation); unit: breaths/min] | 16.52 (2.62)

OUTCOME MEASURES:

1. Primary Outcome: Measurement of AF Cycle Length
Description: Data collected during the study will be used to test an AF cycle length algorithm
Time Frame: One day - day of procedure
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Full Cohort: All enrolled patients
Arm/Group | Full Cohort
Number analyzed (Participants) | 21
ms | 171.64 (27.23)

ADVERSE EVENTS:
Time Frame: Enrollment until hospital discharge, up to 3 days
Arm/Group | Full Cohort
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full Cohort (N=21)
Bleeding from the groin (Vascular disorders) | 1 — The patient had bleeding from the vascular entry site in the groin which required a prolonged hospital stay.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT05477602/Prot_SAP_000.pdf